CLINICAL TRIAL: NCT02606539
Title: Primary Surgery Plus Single Course Methotrexate Versus Primary Methotrexate for Treatment of Gestational Trophoblastic Neoplasms in Low Risk Cases Above 40y: a Randomized Controled Trial
Brief Title: Surgery Plus Single Agent Chemotherapy Versus Primary Chemotherapy for Gestational Trophoblastic Neoplasms
Acronym: SVCGTN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maher elesawi kamel elesawi (Other)
Responsible Party: Sponsor-Investigator, Maher elesawi kamel elesawi, assistant lecturer, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTN and surgery
Record Dates: First submitted 2015-08-08; First posted 2015-11-17 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2015-11

CONDITIONS: Gestational Trophoblastic Neoplasms
Keywords: gestaional trophoblastic neoplasm; hystrectomy; chemotherapy; methotrxate
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — Methotrexate; Surgical Procedures, Operative; Drug Therapy; Leucovorin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery and methotrxate (Active Comparator): The patient will be treated by total abdominal hystrectomy(after written consent laparatomy will be done then pelvic examination for extra uterine spread, palpation of liver, omentum for any gross lesions and then hystrectomt bilateral salpigooophrectomy will be done) plus single course methotrexate(anti folate chemotheraputic agent, vial form given by intramuscular injection) 1mg/kg alternating with calcium folinate 0.1 mg/kg until normalization of B-HCG
  Interventions: Procedure: Total abdominal hysterectomy and methotrexate
- methotrxate (Active Comparator): The patient will be treated by multiple courses of methotrexate( antifolate) 1mg/kg every 14 days each one alternating in every otherday with calcium folinate 0.1 mg/kg till normalization of B-HCG
  Interventions: Drug: Methotrexate plus folinic acid alone

INTERVENTIONS:
Procedure: Total abdominal hysterectomy and methotrexate — After written consent laparotomy will be done then pelvic examination for extra uterine spread, palpation of liver, omentum for any gross lesions and then hystrectomt bilateral salpigooophrectomy will be done) plus single course methotrexate(anti folate chemotheraputic agent, vial form given by intramuscular injection) 1mg/kg every other day alternating with calcium folinate 0.1 mg/kg for 4 doses each cycle then measuring B-HCG (the cycle may be repeated until normalization of B-HCG)
  Other Names: surgery and chemotherapy
  Arms: surgery and methotrxate
Drug: Methotrexate plus folinic acid alone — methotrxate 1mg/kg every other day alternating with calcium folinate 0.1 mg/kg for 4 doses each cycle then measuring B-HCG and cycle repeated until normalization of B-HCG
  Other Names: chemotharapy
  Arms: methotrxate

SUMMARY:
Gestational trophoblastic neoplasm affect women and is sensitive to chemotherapy especially methotrexate and the investigators try to find a role of surgery plus methotrexate instead of multiple doses and cycles of chemotherapy.

DETAILED DESCRIPTION:
Gestational trophoblastic neoplasm affect women and is sensitive to chemotherapy espechialy methotrexate and the investigators try to find a role of surgery plus mehotrexate instead of multiple doses and cycles of chemotherapy that affect the patient quality of life and complication related to both line of management and time of decrease of B-hcg.

ELIGIBILITY:
Inclusion Criteria:

* females
* 40 years or more
* plateau or rising B- hCG titre
* without distant metastasis
* WHO score is less than 7

Exclusion Criteria:

* less than 40 years
* distant metastasis to lung and liver
* chronic medical diseases
* WHO score is more than 7

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
number of primary chemotherapy courses till B-hCG reach less than 5 MU/ML | 1-6 months

SECONDARY OUTCOMES:
quality of life( questionairre) | 1-6 months
  pain scale from zero to 11, return to ordinary activities
complications from management | 1-6 months
  renal, hepatic impairments, anemia,
time interval for B-hCG reach less than 5 MU/ML | 1-6 months
  the time taken for B-hCG to reach below 5 MU/ML

CONTACTS AND LOCATIONS:
Overall Officials: Reda hemida, MD, Principal Investigator — Mansoura University
Locations (2):
- Egypt (2):
  - Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Maher Elesawi Kamel Elesawi, Mīt Ghamr, Eldakahlia